CLINICAL TRIAL: NCT06733545
Title: Study for the Evaluation of the Degree of Skin Satisfaction of Cosmetics Creams PB-011 and PB-012 for Sensitive Skin in Oncological Patients Affected by a Palmoplantar Polyneuropathy Secondary to Chemotherapy or Chemotherapeutic Agents' Fusion to Monoclonal Antibodies (Immunocitostatics)
Brief Title: Study for the Evaluation of the Degree of Skin Satisfaction of a Cosmetic Cream for Sensitive Skin in Oncological Patients Affected by a Palmoplantar Polyneuropathy Secondary to Chemotherapy.
Status: Completed | Type: Observational
Sponsor: PROSPERA BIOTECH S.L. (Industry)
Collaborators: Hospital General Universitario Elche (Other); Hospital Miguel Servet (Other); Hospital del Mar (Other); Hospital Marina Baixa, Alicante (Unknown); Hospital Universitario Ramon y Cajal (Other); Hospital General Universitario Santa Lucia (Other); Hospital Universitari Sagrat Cor, Barcelona (Unknown); Hospital General de Elda (Other); Centre Hospitalier Universitaire Saint Pierre (Other); Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Sponsor
Other Study IDs: 20-PB02
Record Dates: First submitted 2024-11-26; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Quality of Life (QOL); CIPN - Chemotherapy-Induced Peripheral Neuropathy
Keywords: CIPN; Sensitive skin; Quality of life; Chemotherapy; Chemotherapy skin side effects; palmoplantar discomfort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PB-011: Patients starting chemotherapy treatment are given (double blinded) moisturizing cream PB-011 to use once a day in hands. If sensory discomfort appears in hands or feet, the dosage could be increased up to twice a day in hands and feet.
- PB-012: Patients undergoing chemotherapy treatment are given (double blinded) moisturizing cream PB-012 to use once a day in hands. If sensory discomfort appears in hands or feet, the dosage could be increased up to twice a day in hands and feet.

SUMMARY:
It is proposed a controlled research study aimed to evaluating and comparing the degree of skin satisfaction and comfort with cosmetic creams PB-011 and PB-012 in cancer patients who can develop a palmar and plantar peripheral polyneuropathy by treatment with chemotherapy. Both products are cosmetic creams derived from the cosmetic Nocisens® line (for the care of sensitive skin with atopic tendency). The hypothesis that is proposed to test is that the care with PB-011 or PB-012 of the sensitive skin associated with palmar and plantar peripheral polyneuropathy of cancer patients will increase their degree of satisfaction and skin comfort. This study is proposed in patients who are going to start chemotherapeutic treatment. The study conceives two populations: (i) population where PB-011 cream will be tested; and (ii) population that will test PB-012 cream. A sample size of 60 volunteers per population has been estimated to ensure statistical significance. As a qualitative relevant variable for patients, the degree of satisfaction and skin comfort of the volunteers will be assessed by means of questionnaires.

DETAILED DESCRIPTION:
This proof-of-concept clinical trial is a multicenter, double-blind, randomized, placebo-controlled research project approved by the ethics committees of all participating hospitals. Medical oncologists have been responsible for recruiting volunteers, checking that they meet the inclusion and exclusion criteria, obtaining signed informed consent, completing the data collection booklet and collecting the occurrence of CIPN and the degree of CIPN, along with patient follow-up. Once informed consent has been signed, the patients are provided with a PB-011 or the PB-012 formulation and started a daily application on their hands. After the onset of sensory symptoms on hands and/or feet, participants applied the cream twice daily on hands and feet and began responding questionnaires to evaluate the severity of sensorial symptoms.

ELIGIBILITY:
Inclusion Criteria:

* To be older than 18 year old
* To be able to complete questionnaires
* Give informed consent in writing
* Being able to apply the product under test by oneself
* To have been diagnosed with stage I-III primary cancer
* To have received a maximum of one treatment session with chemotherapy (derivatives of taxane, platinum or vincristines)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Life expectancy greater than or equal to 6 months

Exclusion Criteria:

* Not being or having been treated with antidepressants, antiepileptics or HIV medication in the last 3 months
* Pre-existing peripheral neuropathies not related to chemotherapy treatment
* Pre-existing neurodegenerative or neuromuscular disease or history of stroke
* Family history of neuropathic diseases
* Having suffered in the last 6 months: myocardial infarction, unstable angina, stroke, transient ischemic attack, decompensated heart failure requiring hospitalization or class III/IV heart failure.
* Being receiving investigational treatment (being involved in a clinical trial
* Evidence or indication of metastasis affecting the Central Nervous System
* Use of immunosuppressive or immunomodulatory medication that may lead to immunodeficiencies
* Not being treated with topical palmar and/or plantar medication
* Known hypersensitivity to capsaicin
* Having reduced capacity for expression or response to forms
* Not have been under general anesthesia for at least one month before starting the study
* Complication of peripheral polyneuropathy symptoms that require the use of specific medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was anyone over 18 years of age who met the inclusion and exclusion criteria and who was about to start chemotherapy treatment.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Sensory discomfort appearance in hands and/or feet as a measure of quality of life | The estimated period of time over which the event is assessed is up to16 weeks, which correspond from the first CT cycle (cycles are received once a week, 12 CT cycles) up to one month later.
  The appearance of sensory sensations resulting from CIPN will be detected by the oncologists' follow-up. The oncologists will indicate the treatment cycle in which the neuropathy discomfort appears and their degree in the data collection notebook. The study involves following the patient from the first cycle of chemotherapy until one month after the end of treatment.

SECONDARY OUTCOMES:
Skin Discomfort Severity | Questionnaire was done every three weeks until one month after treatment was finished.
  Once recruited volunteers start experiencing sensory skin discomfort in hands/feet and inform their oncologist, a Leonard Scale questionnaire was used to monitor these symptoms (The Leonard Scale1 consists of 14 questions that quantify the subjective intensity of each symptom (e.g. itch, stinging, pain…). Intensity is rated from 1-10, being 1 hardly any and 10 very much).
  1. Leonard GD, Wright MA, Quinn MG, Fioravanti S, Harold N, Schuler B, Thomas RR, Grem JL. Survey of oxaliplatin-associated neurotoxicity using an interview-based questionnaire in patients with metastatic colorectal cancer. BMC Cancer. 2005 Sep 16;5:116. doi: 10.1186/1471-2407-5-116. PMID: 16168057; PMCID: PMC1266024.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Sonia Servitja, Oncologist, Principal Investigator — Servicio de Oncología Médica, Hospital del Mar, 08003 Barcelona (Spain); Maria Castro-Henriques, Oncologist, Principal Investigator — Servicio de Oncología Médica, Hospital del Mar, 08003 Barcelona (Spain); Iñaki Álvarez-Busto, Oncologist, Principal Investigator — Servicio de Oncología Médica, Hospital Universitario Miguel Servet, 50009 Zaragoza (Spain); Maria Asunción Algarra-García, Oncologist, Principal Investigator — Servicio de Oncología Médica, Hospital Marina Baixa, 03570 Villajoyosa, Alicante (Spain); Elena López-Miranda, Oncologist, Principal Investigator — Servicio de Oncología Médica, Hospital Universitario Ramon y Cajal, 28034 Madrid (Spain); Maria I Luengo-Alcázar, Oncologist, Principal Investigator — Servicio de Oncología Médica, Hospital General Universitario Santa Lucía, 30202 Cartagena, Murcia (Spain); Miguel Borregón, Oncologist, Principal Investigator — Servicio de Oncología Médica, Hospital General Universitario de Elche, 03202 Elche, Alicante (Spain); Anna Gassull-Delgado, Nursery, Principal Investigator — Servicio de Oncología Médica, Hospital Universitari Sagrat Cor, 08029 Barcelona (Spain); Ana Gonzaga-López, Oncologist, Principal Investigator — Servicio de Oncología Médica, Hospital General Universitario de Elda, 03600 Elda, Alicante (Spain); Jesus M Poveda-Ferriols, Oncologist, Principal Investigator — CHU St-Pierre-UMC St-Pieter, 1000 Brussels (Belgium)
Locations (1):
- Prospera Biotech,, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data on the anonymised patients such as treatment, number of cycles, sex, age and morbidities during the study could be shared with reviwers or researchers.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: From July of 2022 to July 2027
Access Criteria: Upon request to Prospera Biotech, researchers and doctors will be able to access it. Additional information will be available for peer-reviewers.

REFERENCES:
- [Background] Bae EH, Greenwald MK, Schwartz AG. Chemotherapy-Induced Peripheral Neuropathy: Mechanisms and Therapeutic Avenues. Neurotherapeutics. 2021 Oct;18(4):2384-2396. doi: 10.1007/s13311-021-01142-2. Epub 2021 Oct 21. PMID 34676514
- [Background] Chen X, Gan Y, Au NPB, Ma CHE. Current understanding of the molecular mechanisms of chemotherapy-induced peripheral neuropathy. Front Mol Neurosci. 2024 Apr 10;17:1345811. doi: 10.3389/fnmol.2024.1345811. eCollection 2024. PMID 38660386
- [Background] Aromolaran KA, Goldstein PA. Ion channels and neuronal hyperexcitability in chemotherapy-induced peripheral neuropathy; cause and effect? Mol Pain. 2017 Jan-Dec;13:1744806917714693. doi: 10.1177/1744806917714693. PMID 28580836
- [Background] Nikolaeva-Koleva M, Butron L, Gonzalez-Rodriguez S, Devesa I, Valente P, Serafini M, Genazzani AA, Pirali T, Ballester GF, Fernandez-Carvajal A, Ferrer-Montiel A. A capsaicinoid-based soft drug, AG1529, for attenuating TRPV1-mediated histaminergic and inflammatory sensory neuron excitability. Sci Rep. 2021 Jan 8;11(1):246. doi: 10.1038/s41598-020-80725-z. PMID 33420359
- [Background] Serafini M, Griglio A, Aprile S, Seiti F, Travelli C, Pattarino F, Grosa G, Sorba G, Genazzani AA, Gonzalez-Rodriguez S, Butron L, Devesa I, Fernandez-Carvajal A, Pirali T, Ferrer-Montiel A. Targeting Transient Receptor Potential Vanilloid 1 (TRPV1) Channel Softly: The Discovery of Passerini Adducts as a Topical Treatment for Inflammatory Skin Disorders. J Med Chem. 2018 May 24;61(10):4436-4455. doi: 10.1021/acs.jmedchem.8b00109. Epub 2018 May 15. PMID 29722529
- [Background] Marcotti A, Fernandez-Trillo J, Gonzalez A, Vizcaino-Escoto M, Ros-Arlanzon P, Romero L, Vela JM, Gomis A, Viana F, de la Pena E. TRPA1 modulation by Sigma-1 receptor prevents oxaliplatin-induced painful peripheral neuropathy. Brain. 2023 Feb 13;146(2):475-491. doi: 10.1093/brain/awac273. PMID 35871491
- [Background] Villalba-Riquelme E, de la Torre-Martinez R, Fernandez-Carvajal A, Ferrer-Montiel A. Paclitaxel in vitro reversibly sensitizes the excitability of IB4(-) and IB4(+) sensory neurons from male and female rats. Br J Pharmacol. 2022 Jul;179(14):3693-3710. doi: 10.1111/bph.15809. Epub 2022 Mar 7. PMID 35102580
- [Background] Starobova H, Vetter I. Pathophysiology of Chemotherapy-Induced Peripheral Neuropathy. Front Mol Neurosci. 2017 May 31;10:174. doi: 10.3389/fnmol.2017.00174. eCollection 2017. PMID 28620280
- [Background] Wang DS, Wang ZQ, Chen G, Peng JW, Wang W, Deng YH, Wang FH, Zhang JW, Liang HL, Feng F, Xie CB, Ren C, Jin Y, Shi SM, Fan WH, Lu ZH, Ding PR, Wang F, Xu RH, Li YH. Phase III randomized, placebo-controlled, double-blind study of monosialotetrahexosylganglioside for the prevention of oxaliplatin-induced peripheral neurotoxicity in stage II/III colorectal cancer. Cancer Med. 2020 Jan;9(1):151-159. doi: 10.1002/cam4.2693. Epub 2019 Nov 13. PMID 31724334
- [Background] Gewandter JS, Culakova E, Davis JN, Gada U, Guido JJ, Bearden JD, Burnette B, Shah D, Morrow GR, Mustian K, Sluka KA, Mohile N. Wireless Transcutaneous Electrical Nerve Stimulation (TENS) for Chronic Chemotherapy-Induced Peripheral Neuropathy (CIPN): A Proof-of-Concept Randomized Clinical Trial. J Pain. 2024 May;25(5):104431. doi: 10.1016/j.jpain.2023.11.014. Epub 2023 Nov 21. PMID 37993030
- [Background] Accordino MK, Lee S, Leu CS, Levin B, Trivedi MS, Crew KD, Kalinsky K, Raghunathan R, Faheem K, Harden E, Taboada A, de Oliveira BD, Larson E, Franks L, Honan E, Law C, Hershman DL. Randomized adaptive selection trial of cryotherapy, compression therapy, and placebo to prevent taxane-induced peripheral neuropathy in patients with breast cancer. Breast Cancer Res Treat. 2024 Feb;204(1):49-59. doi: 10.1007/s10549-023-07172-y. Epub 2023 Dec 7. PMID 38060077
- [Background] Mezzanotte JN, Grimm M, Shinde NV, Nolan T, Worthen-Chaudhari L, Williams NO, Lustberg MB. Updates in the Treatment of Chemotherapy-Induced Peripheral Neuropathy. Curr Treat Options Oncol. 2022 Jan;23(1):29-42. doi: 10.1007/s11864-021-00926-0. Epub 2022 Feb 15. PMID 35167004
- [Background] Hershman DL, Lacchetti C, Dworkin RH, Lavoie Smith EM, Bleeker J, Cavaletti G, Chauhan C, Gavin P, Lavino A, Lustberg MB, Paice J, Schneider B, Smith ML, Smith T, Terstriep S, Wagner-Johnston N, Bak K, Loprinzi CL; American Society of Clinical Oncology. Prevention and management of chemotherapy-induced peripheral neuropathy in survivors of adult cancers: American Society of Clinical Oncology clinical practice guideline. J Clin Oncol. 2014 Jun 20;32(18):1941-67. doi: 10.1200/JCO.2013.54.0914. Epub 2014 Apr 14. PMID 24733808
- [Background] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Background] Pachman DR, Qin R, Seisler DK, Smith EM, Beutler AS, Ta LE, Lafky JM, Wagner-Johnston ND, Ruddy KJ, Dakhil S, Staff NP, Grothey A, Loprinzi CL. Clinical Course of Oxaliplatin-Induced Neuropathy: Results From the Randomized Phase III Trial N08CB (Alliance). J Clin Oncol. 2015 Oct 20;33(30):3416-22. doi: 10.1200/JCO.2014.58.8533. Epub 2015 Aug 17. PMID 26282635
- [Background] Burgess J, Ferdousi M, Gosal D, Boon C, Matsumoto K, Marshall A, Mak T, Marshall A, Frank B, Malik RA, Alam U. Chemotherapy-Induced Peripheral Neuropathy: Epidemiology, Pathomechanisms and Treatment. Oncol Ther. 2021 Dec;9(2):385-450. doi: 10.1007/s40487-021-00168-y. Epub 2021 Oct 16. PMID 34655433

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT06733545/Prot_SAP_ICF_000.pdf